CLINICAL TRIAL: NCT03339609
Title: Micturition Reeductation in Children With Cerebral Palsy: Uroflow/EMG Measurement in Healthy Children
Brief Title: Uroflow Measurement With Electromyography (EMG) to Identify Lower Urinary Tract Symptoms (LUTS): Conducted on Healthy Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/766
Record Dates: First submitted 2017-11-06; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Lower Urinary Tract Symptoms; Urologic Diseases
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urologic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate uroflow/EMG testing: Participants performed two direct repetitions of uroflowmetry in combination with EMG.
  Interventions: Diagnostic Test: Uroflow/EMG; Diagnostic Test: US
- uroflow measurement beforehand: Participants performed a preceding measurement of isolated uroflowmetry, followed by two randomized measurements of either isolated uroflowmetry or uroflowmetry with EMG.
  Interventions: Diagnostic Test: Uroflow; Diagnostic Test: Uroflow/EMG; Diagnostic Test: US

INTERVENTIONS:
Diagnostic Test: Uroflow — Isolated uroflow measurement
  Groups: uroflow measurement beforehand
Diagnostic Test: Uroflow/EMG — Uroflow measurement with superficial EMG testing of the pelvic floor
Diagnostic Test: US — Ultrasound of post void residual urine

SUMMARY:
Nowadays there is a growing interest towards non-invasive assessment of urinary dysfunctions in clinical practice. The tendency to use uroflowmetry as a first-line screening tool is based on the inexpensiveness, time efficiency, comfort of the patient, etc. However, it is stated that uroflowmetry as a stand-alone study lacks the potential to make an accurate diagnosis. In regard to this, the International Continence Society indicated that the addition of pelvic floor electromyography might increase the accuracy of this assessment. Despite this recommendation, uroflowmetry in combination with electromyography has not been conducted in a healthy population.

The initial objective of this study was to examine whether adding electromyography to standard uroflowmetry in a healthy paediatric population would change the representation of parameters, especially of voiding patterns. In addition, the influence of several factors on uroflow parameters was analysed to complement current literature.

ELIGIBILITY:
Inclusion Criteria:

• Normal development

Exclusion Criteria:

* (Recurrent) urinary tract infections
* LUTS which interfered with daily life
* Fecal incontinence
* History of genitourinary or renal surgery
* Medication for incontinence during the last 3 months
* Pelvic reeducation during the last 6 months
* Neurologic problems influencing continence

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: continent children with normal development: community sample
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Uroflow curve pattern - Clinical assessment | 2017
  Interpretation by pediatric urologist
Uroflow curve pattern - Mathematical assessment | 2017
  Interpretation using Flow index methodology

SECONDARY OUTCOMES:
Maximal flow | 2017
  Qmax (millilitres/seconds)
post-void residual urine | 2017
  millilitres
voiding time | 2017
  seconds
voided volume | 2017
  millilitres

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No